CLINICAL TRIAL: NCT03059264
Title: Trial Readiness and Endpoint Assessment in Congenital Myotonic Dystrophy
Acronym: TREAT-CDM
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other); University of Western Ontario, Canada, Children's Health Research Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: HM20014211
Record Dates: First submitted 2017-01-25; First posted 2017-02-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Congenital Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CDM: Children with Congenital Myotonic Dystrophy
  Interventions: Other: Natural history
- Control: Healthy Children
  Interventions: Other: Natural history

INTERVENTIONS:
Other: Natural history — Longitudinal disease progression

SUMMARY:
Congenital Myotonic Dystrophy (CDM) is a multi-systemic, dominantly inherited disorder caused by a trinucleotide repeat expansion (CTGn) in the DMPK gene. CDM occurs when the CTGn increases between the adult myotonic dystrophy type-1 (DM1) parent and the child. Children with CDM present at birth with respiratory insufficiency, talipes equinovarus, feeding difficulties and hypotonia. There is a 30% mortality rate in the first year of life. As children grow, they are at risk for intellectual impairment, autistic features, gastrointestinal symptoms, and motor delay.

The investigators will enroll children with CDM between ages 0-15 with visits at baseline and one year to evaluate appropriate physical functional outcomes, cognitive function and quality of life over time. Functional outcome measures will be correlated with potential biomarkers in the children. Completion of these specific aims will extend the understanding of disease progression in CDM and will provide the requisite information for successful therapeutic trials in children with DM.

ELIGIBILITY:
CDM Group

Inclusion Criteria:

* Age 0-15 yrs
* Diagnosis of CDM, based on symptoms and genetic testing of expanded trinucleotide repeats.

Exclusion Criteria:

* Any other non-DM1 illness that would interfere with the ability or results of the study in the opinion of site investigator
* Significant trauma within one month
* Internal metal or devices

Control Group

Inclusion Criteria:

* Age 0-15 yrs
* Healthy children on no medication

Exclusion Criteria:

* Any illness or situation that, in the opinion of the site investigator, has the possibility to interfere with study procedures
* DM type 1 and 2

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study proposes a longitudinal evaluation of 100 children with CDM and 50 healthy controls, stratified into the following age cohorts: 0-2 years, 11 months; 3 years to 6 years, 11 months; and 7 years and older. The age cohorts are created to ensure an even distribution across all ages.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Grip Strength | 1 year
  Measure of force generated by hand grip

SECONDARY OUTCOMES:
Congenital and Childhood Onset Myotonic Dystrophy Health Index (CCMDHI) | 1 year
  Disease specific patient and parent reported outcome measure of quality of life
6-minute walk | 1 year
  Assess distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance
Behavior Rating Inventory of Executive Function (BRIEF) | 1 year
  An 86-item parent/caregiver-proxy and teacher-proxy rating form of executive function skills in every-day settings such as school, home, and social situations
Lip Force | 1 year
  Measure of force generation by orbicularis oris

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (3):
- Virginia Commonwealth University, Richmond, Virginia, United States
- Pediatric Neuromuscular Research, Children's Hospital - LHSC, London, Ontario, Canada
- Centro Clinico Nemo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No